CLINICAL TRIAL: NCT02378506
Title: A Single-arm, Open-label Study To Assess The Immunogenicity, Safety, And Efficacy Of Etanercept Manufactured Using The High Capacity Process Administered To Subjects With Rheumatoid Arthritis
Brief Title: Study to Assess the Immunogenicity, Safety, and Efficacy of High Capacity Process Etanercept in Rheumatoid Arthritis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1801359; 2013-004569-16 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-03-04 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ETN 50mg QW (Experimental)
  Interventions: Biological: etanercept

INTERVENTIONS:
Biological: etanercept — 50mg subcutaneous, once weekly, 24 weeks

SUMMARY:
Open-label immunogenicity, safety and efficacy study of etanercept manufactured using the high capacity process. Descriptive results will be provided however a formal hypothesis will not be tested in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active disease with presence of at least 4 tender joints and 4 swollen joints.
* Either the patient or a designee must be capable of administering the subcutaneous injection of study drug.

Exclusion Criteria:

* Prior treatment with etanercept.
* Presence of active infection or active or untreated tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- Bulgaria (4):
  - MHAT Plovdiv, Plovdiv
  - DCC "Aleksandrovska" EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski" EAD, Sofia, Sofia
  - Medical Center - "New rehabilitation center" EOOD, Stara Zagora
- Croatia (2):
  - Chc Rijeka, Rijeka
  - Medicinski Centar Kuna Peric, Zagreb
- Germany (5):
  - Centrum für innovative Diagnostik und Therapie, Frankfurt am Main, Hesse
  - Rheumaforschung - Studienambulanz Dr. Wassenberg, Ratingen, North Rhine-Westphalia
  - Schlosspark-Klinik, Innere Medizin II, Rheumatologie, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Immunologisches Zentrum Vogelsang-Gommern GmbH, Vogelsang-Gommern
- Greece (3):
  - Rheumatology Department, Rion Patras, Achaia
  - University Hospital of Heraklion, Heraklion, Crete
  - Rheumatology Unit, Thessaloniki
- Hungary (3):
  - Qualiclinic Kft., Budapest
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Szabolcs-Szatmar-Bereg megyei, Nyíregyháza
- Poland (4):
  - Krakowskie Centrum Medyczne sp. Z.O.O, Krakow
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn
  - Prywatna Praktyka Lekarska Prof. UM dr hab.med. Pawel Hrycaj, Poznan
  - Reumatika-Centrum Reumatologii, Warsaw
- Institute of Rheumatology, Belgrade, Beograd, Serbia
- Slovakia (6):
  - Reumatologicka ambulancia, Bratislava
  - AAGS, s.r.o., Dunajská Streda
  - Reumatologicka ambulancia, MUDr. Zuzana Cizmarikova, s.r.o., Poprad
  - REUMEX s.r.o., Rimavská Sobota
  - REUMA-GLOBAL s.r.o., Trnava
  - Reumatologicka ambulancia, Žilina
- South Africa (3):
  - Panorama Medical Centre, Panorama, Cape Town
  - Wits Clinical Research CMJAH Clinical Trial Site, Parktown, Johannesburg
  - St. Augustines Hospital, Durban/Berea, KwaZulu-Natal

REFERENCES:
- [Derived] Polak P, Peric P, Louw I, Gaylord SM, Williams T, Becker JC, Pedersen R, Korth-Bradley J, Vlahos B. A single-arm, open-label study to assess the immunogenicity, safety, and efficacy of etanercept manufactured using the serum-free, high-capacity manufacturing process administered to patients with rheumatoid arthritis. Eur J Rheumatol. 2019 Jan;6(1):23-28. doi: 10.5152/eurjrheum.2018.18078. PMID 30451655
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801359&StudyName=Study%20to%20Assess%20the%20Immunogenicity%2C%20Safety%2C%20and%20Efficacy%20of%20Etanercept%20Manufactured%20Using%20the%20High%20Capacity%20Process%20Administered%20to%20Rh

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants with moderate to severe rheumatoid arthritis, received subcutaneous Etanercept 50 milligram (mg) once weekly up to Week 24 and were followed up to Week 28.
Period: Overall Study
Arm/Group | Etanercept
Started | 188
Treated | 187
Completed | 163
Not Completed | 25
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 2
Not completed — Death | 1
Not completed — Adverse Event | 14
Not completed — Randomized But Not Treated | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Arm/Group | Etanercept
Number analyzed (Participants) | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Positive Etanercept Anti-Drug Antibody (ADA) Status at Week 12
Description: Participants who developed anti-drug antibodies after treatment with Etanercept were evaluated. Percentage of participants with positive Etanercept anti-drug antibodies were summarized.
Time Frame: Week 12
Population: Analysis set included all participants who had taken at least 1 dose of study medication and had at least 1 Etanercept anti-drug antibody evaluation. Here, "Number of Participants Analyzed" (N) signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 158
percentage of participants | 1.9 [0.5 to 5.0]

2. Primary Outcome: Percentage of Participants With Positive Etanercept Anti-Drug Antibody Status at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Analysis set included all participants who had taken at least 1 dose of study medication and had at least 1 Etanercept anti-drug antibody evaluation. Here, "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 175
percentage of participants | 2.9 [1.1 to 6.1]

3. Secondary Outcome: Percentage of Participants With Positive Etanercept Neutralizing Anti-Drug Antibody Status: Throughout Study Treatment
Description: Percentage of participants with positive Etanercept neutralizing anti-drug antibodies were summarized.
Time Frame: Baseline (Day 1) up to Week 24
Population: Analysis set included all participants who had taken at least 1 dose of study medication and had at least 1 Etanercept anti-drug antibody evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 176
percentage of participants | 0.00 [0.00 to 1.4]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to Week 28 (Follow-up)
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 187
participants
  AEs | 90
  SAEs | 9

5. Secondary Outcome: Number of Participants With Investigator-Identified Serious Infections
Description: Infection was considered as serious by investigator for any of the following outcomes: death; life-threatening; required initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity or congenital anomaly/birth defect.
Time Frame: Baseline (Day 1) up to Week 28 (Follow-up)
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 187
participants | 3

6. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions included injection site erythema, swelling, pain and warmth.
Time Frame: Baseline (Day 1) up to Week 28 (Follow-up)
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 187
participants | 27

7. Secondary Outcome: Number of Participants With Grade 3 and 4 Clinical Laboratory Abnormalities
Description: Laboratory abnormalities(national cancer institute toxicity criteria version 4.0),Grade 3:neutrophil (greater than or equal to[>=]0.5,less than[<]1.0 10^9/L),lymphocyte (<0.5 10^9/L),hemoglobin (Hb) (<80,>=65 gram per liter [g/L]),platelet(<50.0,>=25.0 10^9/L),white blood count(WBC) (<2.0, >=1.0 10^9/L);alkaline phosphatase (AP),aspartate aminotransferase(AST),alanine aminotransferase(ALT) (greater than[>]5.0*upper range [UR], <=20.0*UR unit per liter[U/L]);bilirubin(>1.5*UR, less than or equal to[<=]3.0*UR micromole per liter[mcmol/L]);creatinine(>3.0*UR, <=6.0*UR mcmol/L);albumin (<20.0 g/L),urea(>3.0*UR, <=4.0*UR g/L);potassium (K)-high,low (>6.0,<=7.0or<3.0,>=2.5 mcmol/L); sodium(Na)-high,low(>155, <=160 or <130, >=120 mcmol/L)and Grade 4: neutrophil(<0.5 10^9/L),Hb (<65 g/L);platelet (<25.0 10^9/L); WBC(<1.0 10^9/L);AP,AST,ALT(>20.0*UR U/L);bilirubin(>3.0*UR mcmol/L);creatinine (>6.0*UR mcmol/L);urea (>4.0*UR g/L);K-high,low (>7.0or<2.5 mcmol/L);Na-high, low (>160or<120 mcmol/L).
Time Frame: Baseline (Day 1) up to Week 28 (Follow-up)
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 187
participants | 5

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 responder: participants with 20 percent (%) improvement in tender and swollen 28-joint counts and 20% improvement in at least 3 of the 5 measures: participant global assessment of arthritis (PtGA), physician global assessment of arthritis (PGA), participant pain visual analogue scale (Pain-VAS), health assessment questionnaire-disability index (HAQ-DI) and C-reactive protein. PtGA: participant assessed overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. PGA: physician judged participant's overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. Pain-VAS: participant assessed arthritis pain by 100 millimeter (mm) VAS, score: 0 mm (no pain) to 100 mm (extreme pain), higher score=more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score=more disability. Percentage of participants with ACR20 response were reported.
Time Frame: Week 4, 12, 24
Population: Modified intent-to-treat (mITT) population included all participants who had taken at least 1 dose of study medication. Here, "n" signifies number of participants who were evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 187
percentage of participants
  Week 4 (n =186) | 55.9 [48.7 to 62.9]
  Week 12 (n =179) | 76.5 [69.9 to 82.3]
  Week 24 (n =161) | 82.0 [75.5 to 87.3]

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 responder: participants with 50% improvement in tender and swollen 28-joint counts and 50% improvement in at least 3 of the 5 measures: participant global assessment of arthritis (PtGA), physician global assessment of arthritis (PGA), participant pain visual analogue scale (Pain-VAS), health assessment questionnaire-disability index (HAQ-DI) and C-reactive protein. PtGA: participant assessed overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. PGA: physician judged participant's overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. Pain-VAS: participant assessed arthritis pain by 100 millimeter (mm) VAS, score: 0 mm (no pain) to 100 mm (extreme pain), higher score=more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score=more disability. Percentage of participants with ACR50 response were reported.
Time Frame: Week 4, 12, 24
Population: mITT population included all participants who had taken at least 1 dose of study medication. Here, "n" signifies number of participants who were evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 187
percentage of participants
  Week 4 (n =186) | 16.1 [11.4 to 21.9]
  Week 12 (n =179) | 36.3 [29.5 to 43.5]
  Week 24 (n =161) | 57.8 [50.1 to 65.2]

10. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 responder: participants with 70% improvement in tender and swollen 28-joint counts and 70% improvement in at least 3 of the 5 measures: participant global assessment of arthritis (PtGA), physician global assessment of arthritis (PGA), participant pain visual analogue scale (Pain-VAS), health assessment questionnaire-disability index (HAQ-DI) and C-reactive protein. PtGA: participant assessed overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. PGA: physician judged participant's overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. Pain-VAS: participant assessed arthritis pain by 100 millimeter (mm) VAS, score: 0 mm (no pain) to 100 mm (extreme pain), higher score=more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score=more disability. Percentage of participants with ACR70 response were reported.
Time Frame: Week 4, 12, 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 187
percentage of participants
  Week 4 (n =186) | 3.2 [1.4 to 6.5]
  Week 12 (n =179) | 13.4 [9.0 to 19.0]
  Week 24 (n =161) | 26.7 [20.3 to 33.9]

11. Secondary Outcome: Change From Baseline in Disease Activity Scale Based on 28 Joint Count Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Week 4, 12 and 24
Description: DAS28: measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from number of swollen joints (SJC) and tender joints (TJC ) using the 28 joints count, erythrocyte sedimentation rate (millimeter per hour [mm/hour]) and participant's general health visual analog scale assessment (scores: 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (ESR) score: 0 (none) to 10 (extreme disease activity), higher scores indicate more disease activity. DAS28-4 (ESR) less than (<) 2.6= remission, <3.2= low disease activity, greater than or equal to (>=) 3.2 to 5.1= moderate disease activity and >5.1= high disease activity.
Time Frame: Baseline, Week 4, 12, 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 187
units on a scale
  Baseline (n =187) | 6.2 (0.93)
  Change at Week 4 (n =186) | -1.5 (1.04)
  Change at Week 12 (n =180) | -2.3 (1.19)
  Change at Week 24 (n =162) | -2.8 (1.27)

12. Secondary Outcome: Change From Baseline in Disease Activity Scale Based on 28 Joint Count C-Reactive Protein (4 Variables) (DAS28-4 [CRP]) at Week 4, 12 and 24
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated from the number of swollen joints and tender joints using the 28 joints count, C-Reactive protein (milligram per liter [mg/L]) and participant's general health visual analog scale assessment (scores ranging 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (CRP) score range: 0 (none) to 10 (extreme disease activity), higher scores indicate more disease activity. DAS28-4 (CRP) less than (<) 2.6= remission, <3.2= low disease activity, greater than or equal to (>=) 3.2 to 5.1= moderate disease activity and >5.1= high disease activity.
Time Frame: Baseline, Week 4, 12, 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 187
units on a scale
  Baseline (n =187) | 5.4 (0.91)
  Change at Week 4 (n =187) | -1.5 (1.02)
  Change at Week 12 (n =179) | -2.2 (1.09)
  Change at Week 24 (n =162) | -2.5 (1.17)

13. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 4, 12 and 24
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each item scored on 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: Baseline, Week 4, 12, 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 187
units on a scale
  Baseline (n =186) | 1.3 (0.58)
  Change at Week 4 (n =186) | -0.3 (0.39)
  Change at Week 12 (n =179) | -0.4 (0.48)
  Change at Week 24 (n =161) | -0.5 (0.56)

14. Primary Outcome: Percentage of Participants With Positive Etanercept Anti-Drug Antibody Status: Throughout Study Treatment
Description: as for outcome 1
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 176
percentage of participants | 4.5 [2.2 to 8.4]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Week 28 (follow-up)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 9/187
Other Adverse Events (participants affected / at risk) | 85/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=187)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Major depression (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Etanercept (N=187)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Retinal detachment (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Influenza like illness (General disorders) | 1
Injection site erythema (General disorders) | 20
Injection site nodule (General disorders) | 1
Injection site pruritus (General disorders) | 7
Injection site rash (General disorders) | 2
Injection site reaction (General disorders) | 5
Injection site swelling (General disorders) | 3
Injection site urticaria (General disorders) | 1
Injection site vesicles (General disorders) | 1
Malaise (General disorders) | 1
Peripheral swelling (General disorders) | 1
Hepatic cyst (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Asymptomatic bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Genitourinary tract infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 13
Otitis media acute (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 13
Urinary tract infection (Infections and infestations) | 4
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood pressure diastolic abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Migraine (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Impulsive behaviour (Psychiatric disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1/159 — This event was gender specific.
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.